CLINICAL TRIAL: NCT02988375
Title: Sleep to Prevent Evolving Affecting Disorders
Acronym: SPREAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Christopher Drake, Director of Sleep Research, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10320
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Insomnia, Primary; Depression
Keywords: insomnia; depression; digital CBTI; online CBTI
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dCBTI (Experimental): Online access to the digital CBTI program Sleepio
  Interventions: Behavioral: dCBTI
- Sleep Education (Placebo Comparator): Weekly email messages with sleep hygiene recommendations
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: dCBTI
  Arms: dCBTI
Behavioral: Sleep Education
  Arms: Sleep Education

SUMMARY:
The primary objective of the proposed research is to determine the efficacy of Digital Cognitive Behavior Therapy (dCBTI) in reducing severity of depression and also in preventing the incidence and relapse of depression among insomniacs. In addition, we will identify salient sociological/environmental variables, such as age, sex, education, socioeconomic status (SES), racial/ethnic minority-status, work schedule, child-care responsibilities (i.e., having children under the age of 3), stigma, that moderate the effects of this intervention.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of Digital Cognitive Behavior Therapy for Insomnia (dCBTI) in reducing severity of depression and also in preventing the incidence and relapse of depression among insomniacs. dCBTI is an online form of Cognitive Behavioral Therapy (CBT) used with people who experience trouble sleeping at night (insomniacs). This study will allow us to determine whether this form of digital therapy is helpful in reducing the severity of depression and in preventing the development and relapse of depression in people suffering from insomnia.

Participants will be recruited from several well-developed sources, including the HFHS Sleep Center Clinical database. Once a participant meets inclusion criteria and provides consent, a link to the internet portal will be provided to complete the remaining survey questions. After completion of this assessment, participants will be automatically randomized to one of 2 active online insomnia treatment conditions. Each treatment involves 6 weekly "sessions" which each take up to 20 minutes to complete.

A post-treatment questionnaire immediately following the 6-week treatment phase will be completed. In addition, a follow up questionnaire assessment will be completed approximately 1 year after treatment. Each of the 3 separate questionnaires will take 20-30 minutes to complete. Participants will be compensated.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition(DSMV) criteria for insomnia

Exclusion Criteria:

* Lack of insomnia, untreated sleep disorder (e.g., obstructive sleep apnea, restless leg syndrome), bipolar disorder, history of seizure disorder, high depression chronicity (self-reported daily or near daily depressed mood and anhedonia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1385 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Drake, PhD, Principal Investigator — Henry Ford Medical Center - Columbus
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheng P, Kalmbach DA, Hsieh HF, Castelan AC, Sagong C, Drake CL. Improved resilience following digital cognitive behavioral therapy for insomnia protects against insomnia and depression one year later. Psychol Med. 2023 Jul;53(9):3826-3836. doi: 10.1017/S0033291722000472. Epub 2022 Mar 8. PMID 35257648
- [Derived] Cheng P, Casement MD, Cuellar R, Johnson DA, Kalmbach D, Cuamatzi Castelan A, Drake CL. Sleepless in COVID-19: racial disparities during the pandemic as a consequence of structural inequity. Sleep. 2022 Jan 11;45(1):zsab242. doi: 10.1093/sleep/zsab242. PMID 34788453
- [Derived] Cheng P, Casement MD, Kalmbach DA, Castelan AC, Drake CL. Digital cognitive behavioral therapy for insomnia promotes later health resilience during the coronavirus disease 19 (COVID-19) pandemic. Sleep. 2021 Apr 9;44(4):zsaa258. doi: 10.1093/sleep/zsaa258. PMID 33249492
- [Derived] Cheng P, Kalmbach DA, Tallent G, Joseph CL, Espie CA, Drake CL. Depression prevention via digital cognitive behavioral therapy for insomnia: a randomized controlled trial. Sleep. 2019 Oct 9;42(10):zsz150. doi: 10.1093/sleep/zsz150. PMID 31535688

RESULTS

PARTICIPANT FLOW:
Groups:
- dCBTI: Online access to the digital CBTI program Sleepio
  dCBTI
- Sleep Education: Weekly email messages with sleep hygiene recommendations
  Sleep Education
Period: Overall Study
Arm/Group | dCBTI | Sleep Education
Started | 946 | 439
Completed | 358 (non-completed subjects consist entirely of participants who were randomized, but failed to initiate the treatment or who stopped doing the dcbti treatment prior to completion of the study.) | 300 (non-completed subjects consist entirely of participants who were randomized, but failed to initiate the treatment or who stopped doing the control treatment prior to completion of the study.)
Not Completed | 588 | 139

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | dCBTI | Sleep Education | Total
Number analyzed (Participants) | 946 | 439 | 1385
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 853 | 376 | 1229
  >=65 years | 93 | 63 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (15.8) | 45.7 (15.1) | 45 (1.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 737 | 351 | 1088
  Male | 209 | 88 | 297
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 16 | 8 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 171 | 109 | 280
  White | 710 | 294 | 1004
  More than one race | 15 | 9 | 24
  Unknown or Not Reported | 31 | 16 | 47

OUTCOME MEASURES:

1. Primary Outcome: Severity of Depression as Measured by the Quick Inventory of Depressive Symptomatology (QIDS) Pre-Treatment
Description: Severity of depression as measured by the Quick Inventory of Depressive Symptomatology (QIDS; ranges 0-27 with higher scores meaning greater severity) and incidence of depression
Time Frame: Pre-treatment (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | dCBTI | Sleep Education
Number analyzed (Participants) | 358 | 300
score on a scale | 10.8 (4.5) | 10.8 (4.6)

2. Primary Outcome: Severity of Depression as Measured by the Quick Inventory of Depressive Symptomatology (QIDS) Post-Treatment
Description: Severity of depression as measured by the Quick Inventory of Depressive Symptomatology (QIDS; ranges 0-27 with higher scores meaning greater severity)
Time Frame: Post-treatment (~6 week after Screening)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | dCBTI | Sleep Education
Number analyzed (Participants) | 358 | 300
score on a scale | 3.9 (4.0) | 6.4 (4.2)

3. Primary Outcome: Severity of Depression as Measured by the Quick Inventory of Depressive Symptomatology (QIDS), 1-year Follow-up
Description: as for outcome 2
Time Frame: 1-year follow-up (58 week after screening)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | dCBTI | Sleep Education
Number analyzed (Participants) | 326 | 283
score on a scale | 4.7 (4.3) | 6.5 (4.3)

4. Primary Outcome: Severity of Symptoms of Insomnia [Time Frame: Pre-treatment (Day 1)]
Description: Insomnia Severity Index Score (ISI; total score range 0-28, with higher scores meaning greater severity)
Time Frame: Pre-treatment (Day 1)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | dCBTI | Sleep Education
Number analyzed (Participants) | 358 | 300
score on a scale | 17.8 (4.2) | 17.7 (4.3)

5. Secondary Outcome: Severity of Symptoms of Insomnia - Post Treatment
Description: Insomnia Severity Index Score (ISI; total score range 0-28, with higher scores meaning greater severity)
Time Frame: Post-treatment (~6 week after Screening)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | dCBTI | Sleep Education
Number analyzed (Participants) | 358 | 300
score on a scale | 17.9 (4.3) | 17.7 (4.4)

6. Secondary Outcome: Severity of Symptoms of Insomnia - 1 Year Post Treatment
Description: Insomnia Severity Index Score (ISI; total score range 0-28, with higher scores meaning greater severity)
Time Frame: 1-year follow-up (58 week after screening)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | dCBTI | Sleep Education
Number analyzed (Participants) | 326 | 283
score on a scale | 8.2 (6.2) | 12.8 (5.6)

ADVERSE EVENTS:
Time Frame: AE not reported.
Description: The definition of adverse event and/or serious adverse event doesn't differ from the clinicaltrials.gov.
Arm/Group | dCBTI | Sleep Education
All-Cause Mortality (participants affected / at risk) | 0/946 | 0/439
Serious Adverse Events (participants affected / at risk) | 0/946 | 0/439
Other Adverse Events (participants affected / at risk) | 0/946 | 0/439

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT02988375/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT02988375/ICF_001.pdf